CLINICAL TRIAL: NCT05255263
Title: Programmed Intermittent Epidural Bolus vs. Continuous Epidural Infusion: a Multicenter, Pragmatic, Cluster-randomized Trial
Brief Title: Goal-directed Labor Epidural Analgesia Maintenance
Acronym: GLEAM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is currently on hold, pending further evaluation and coordination.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GLEAM
Record Dates: First submitted 2021-12-06; First posted 2022-02-24 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Labor Onset and Length Abnormalities
Keywords: Cesarean Delivery; Programmed Intermittent Epidural Bolus (PIEB); Continuous Epidural Infusion (CEI); Patient-Controlled Epidural Analgesia (PCEA); Normal Spontaneous Vaginal Delivery (NSVD); Instrumental Vaginal Delivery; Second Stage of Labor

STUDY DESIGN:
Intervention Model Description: Pragmatic, cluster-randomized, open-labeled, multiple-crossover trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Programmed Intermittent Epidural Bolus (Active Comparator): Intermittent epidural bolus as the first line labor epidural analgesia maintenance infusion
  Interventions: Other: PIEB
- Continuous Epidural Infusion (Active Comparator): Continuous epidural infusion as the first line labor epidural analgesia maintenance infusion
  Interventions: Other: CEI

INTERVENTIONS:
Other: PIEB — Programmed Intermittent Epidural Bolus with Patient-Controlled Epidural Analgesia
  Arms: Programmed Intermittent Epidural Bolus
Other: CEI — Continuous Epidural Infusion with Patient-Controlled Epidural Analgesia
  Arms: Continuous Epidural Infusion

SUMMARY:
The GLEAM trial is a multicenter, pragmatic, cluster-randomized trial to assess the effects of programmed intermittent epidural bolus versus continuous epidural infusion on the rate of spontaneous vaginal delivery and several other clinically-relevant outcomes.

DETAILED DESCRIPTION:
BACKGROUND: The goal of Labor Epidural Analgesia (LEA) to provide optimal analgesia while limiting any impact on the course of labor. Until recently, the most common technique for epidural analgesia was a combination of continuous epidural infusion (CEI) and patient controlled epidural analgesia (PCEA). CEI delivers an infusion of local anesthetic into the epidural space at a constant rate. Programmed intermittent epidural bolus (PIEB)-a more recently-developed alternative to CEI-delivers intermittent boluses of local anesthetic into the epidural space at scheduled time intervals.

A series of randomized control trials (RCT) have compared PIEB and CEI with overall results favoring PIEB for superior analgesia. However, CEI has been shown to be associated with an increased amount of local anesthetic consumption, which may increase the degree of motor blockade, placing parturients at higher risk for instrumental and cesarean deliveries. Studies to date have offered conflicting conclusions on whether CEI is associated with a reduced rates of normal spontaneous vaginal delivery (NSVD).

AIM: The GLEAM trial aims to investigate the hypothesis that PIEB will have higher rates of NSVD than CEI. The effects of CEI vs. PIEB on cesarean delivery rate, instrumental vaginal delivery rate, length of second stage of labor, failed epidural rate.

TRIAL DESIGN: Multi-center, pragmatic, cluster-randomized trial

* Centers will be assigned to use either PIEB or CEI for the first-line labor epidural analgesia maintenance infusion for clusters of minimum one month duration
* Participating institutions will be recruited via the Society for Obstetric Anesthesia and Perinatology (SOAP) Research Network
* Centers must use an epidural solution with a low concentration of local anesthesia with an opioid.
* Both PIEB and CEI must include PCEA - rates and volumes are determined by the institution
* Neuraxial anesthesia can be initiated with Dural Puncture Epidural (DPE), Combined Spinal Epidural (CSE) or epidural bolus
* Our sample will consist of all women, at least 18 years of age, who were admitted to the labour & delivery ward for planned vaginal delivery and had neuraxial analgesia
* Data will be collected in routine clinical care and automatically extracted from the electronic health record (EHR)

PARTICIPATING SITE CRITERIA:

* Routinely provided LEA with Ropivacaine ≤ 0.125% or Bupivacaine ≤ 0.1% epidural solutions with fentanyl (1-3 mcg/ml)
* Can provide LEA with PIEB or CEI
* Must include PCEA as part of all LEA regardless of PIEB or CEI

ELIGIBILITY:
Inclusion Criteria:

* Requests labor epidural analgesia requiring epidural maintenance with local anesthesia and opioid for planned vaginal delivery

Exclusion Criteria:

* Planned cesarean delivery
* Planned operative vaginal delivery
* Epidural time (placement to delivery) < 1 hour

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Spontaneous Vaginal Delivery | Delivery
  Rate of Spontaneous Vaginal Delivery (Percent of total deliveries)

SECONDARY OUTCOMES:
Cesarean Delivery | Delivery
  Rate of Cesarean Delivery (Percent of total deliveries)
Instrumental Vaginal Delivery | Delivery
  Rate of Instrumental Vaginal Delivery (Percent of total deliveries)
Length of Second Stage | During labor up to time of delivery
  Length of Second Stage of Labor (hours)
Failed Epidural | During labor up to time of delivery
  Rate of Failed Epidural, requiring general anesthesia or epidural replacement. (Percent of total labor epidural anesthetics)
Local anesthetic concentration | During labor up to time of delivery
  Local anesthetic concentration (Percent solution)
Epidural opioids used | During labor up to time of delivery
  Epidural opioid (identity of opioid)
Epidural opioids used | During labor up to time of delivery
  Epidural opioid concentration (µg/mL)
CEI rate | During labor up to time of delivery
  Continuous Epidural Infusion Rate (mL/hr)
PIEB Volume | During labor up to time of delivery
  Programmed Intermittent Epidural Bolus Volume (mL)
PIEB Interval | During labor up to time of delivery
  Programmed Intermittent Epidural Bolus (minutes)
PCEA Volume | During labor up to time of delivery
  Patient-Controlled Epidural Analgesia bolus volume (mL)
PCEA Lockout | During labor up to time of delivery
  Patient-Controlled Epidural Analgesia lockout time (minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Xu J, Zhou J, Xiao H, Pan S, Liu J, Shang Y, Yao S. A Systematic Review and Meta-Analysis Comparing Programmed Intermittent Bolus and Continuous Infusion as the Background Infusion for Parturient-Controlled Epidural Analgesia. Sci Rep. 2019 Feb 22;9(1):2583. doi: 10.1038/s41598-019-39248-5. PMID 30796286
- [Background] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Background] McKenzie CP, Cobb B, Riley ET, Carvalho B. Programmed intermittent epidural boluses for maintenance of labor analgesia: an impact study. Int J Obstet Anesth. 2016 May;26:32-8. doi: 10.1016/j.ijoa.2015.11.005. Epub 2015 Nov 27. PMID 26775896
- [Background] Tien M, Allen TK, Mauritz A, Habib AS. A retrospective comparison of programmed intermittent epidural bolus with continuous epidural infusion for maintenance of labor analgesia. Curr Med Res Opin. 2016 Aug;32(8):1435-40. doi: 10.1080/03007995.2016.1181619. Epub 2016 May 20. PMID 27100210
- [Background] Onuoha OC. Epidural Analgesia for Labor: Continuous Infusion Versus Programmed Intermittent Bolus. Anesthesiol Clin. 2017 Mar;35(1):1-14. doi: 10.1016/j.anclin.2016.09.003. Epub 2016 Dec 12. PMID 28131113